CLINICAL TRIAL: NCT06776614
Title: A Comparative-effectiveness Study on Expansion Craniotomy Versus Decompressive Craniectomy for Surgical Management of Traumatic Brain Injury in Patients With Intracranial Compartment Syndrome
Brief Title: Effectiveness of Surgical Procedures for Acute Cranial Expansion in Traumatic Brain Injury
Acronym: E-SPACE-TBI
Status: Not yet recruiting | Type: Observational
Sponsor: Meditech Foundation (Other)
Responsible Party: Principal Investigator, Andres M. Rubiano, Principal Investigator, Meditech Foundation
Other Study IDs: CEIM-2024-12-102
Record Dates: First submitted 2025-01-07; First posted 2025-01-15 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-01

CONDITIONS: Traumatic Brain Injuries; Intracranial Hypertension
Keywords: Traumatic Brain Injury; Intracranial Compartment Syndrome; Decompressive Craniectomy; Expansive Craniotomy
MeSH Terms: conditions — Brain Injuries, Traumatic; Intracranial Hypertension | interventions — Decompressive Craniectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Decompressive Craniectomy Group: Patients with early emergency room (ER) diagnosis of intracranial compartment syndrome who underwent a classical hemicranial decompressive craniectomy procedure
  Interventions: Procedure: Decompressive Craniectomy
- Expansion Craniotomy Group: Patients with early ER diagnosis of intracranial compartment syndrome underwent a specific decompressive craniectomy procedure called expansion craniotomy, with fixation of the bone graft 1cm over the external table of the skull with a set of specific mini plates (Rialto System).
  Interventions: Procedure: Expansion Craniotomy

INTERVENTIONS:
Procedure: Decompressive Craniectomy — The DC will be performed through a standard trauma incision, a retro-auricular "C-shape" or a "Kempe" incision and execute a 15x15 cm craniotomy with a "C-shape" durotomy. Dural closure will be at the discretion of the surgeon and the availability of resources, including duroplasty with aponeurotic galea, a suturable dural patch, a non-suturable dural patch, or simply a superficial dural cover with hemostatic materials like Surgicel® or Gelfoam®. There are multiple techniques for DC. The elected technique will be at the discretion of the treating neurosurgeon, but only front-parietal-temporal DC will be considered. The removed bone flap may be stored in an abdominal pouch in the right or left upper abdominal quadrants or by freezing in a bone or blood bank freezer.
  Other Names: Cranial Decompression; Hemi Craniectomy
  Groups: Decompressive Craniectomy Group
Procedure: Expansion Craniotomy — The EC will be performed through a retro-auricular "C-shape" incision and executing a 15x15 cm craniotomy with a "C-shape" durotomy. Dural closure will be at the discretion of the surgeon and the availability of resources, including duroplasty with aponeurotic galea, a suturable dural patch, a non-suturable dural patch, or simply a superficial dural cover with hemostatic materials like Surgicel® or Gelfoam®. The expansion craniotomy will be finished with a cranioplasty using a full set of 3-5 "Rialto" plates for bone graft closure. The selected technique will be at the discretion of the treating neurosurgeon, but only front-parietal-temporal EC will be considered.
  Other Names: Hinge Craniotomy
  Groups: Expansion Craniotomy Group

SUMMARY:
Traumatic brain injury (TBI) patients often exhibit an increase in their intracranial volume due to blood collection or brain tissue edema. When the volume of any intracranial compartment exceeds a critical threshold, the compensatory mechanisms become exhausted, compromising intracranial compliance and blood supply, which leads to intracranial compartment syndrome (ICCS). The presence of this condition exacerbates brain damage through secondary injury. When less invasive measures to counteract ICCS prove to be insufficient, cranial decompression is recommended, with decompressive craniectomy (DC) being the preferred technique.

Although its effectiveness has been demonstrated, DC is also associated with an incidence of complications. Expansive craniotomy (EC) has been proposed as an alternative that can increase the benefits of cranial decompression provided by DC while reducing the associated complications. This observational study will compare the functional outcomes and complications of patients managed by DC and EC.

DETAILED DESCRIPTION:
In cranial decompression, a cranial vault bone graft is removed and left out to be stored in a bone bank or an abdominal pouch generated during the surgery. In the cranial expansion, the cranial vault bone graft is fixed in an elevated position 1 - 1.5 cm above the external cranial table and fixed by 3-5 metallic plates placed during surgery.

Participants' progress will be observed during their hospital stay and assessed for 1 year through structured telephone follow-ups. The main outcomes will include functional recovery and the rate of complications such as operative site infections, and/or reinterventions. By comparing these two surgical methods, the study seeks to determine whether the expansion craniotomy improves outcomes for TBI patients while maintaining or enhancing the safety and reliability of the cranial decompression procedure.

Currently, decompressive craniectomy (DC) is the most frequently used technique. The Brain Trauma Foundation's current guidelines discuss it and describe the actual evidence. This technique will serve as a comparator for expansion craniotomy (EC). The allocation of patients to the intervention will be based on the clinical criteria of the treating neurosurgeon as long as the patients meet the inclusion criteria and do not present any exclusion criteria.

Neurosurgeons will describe the reason(s) why one technique or another was indicated and why the surgical approach was selected. The EC technique is standardized and will be performed through a retro-auricular "C-shape" incision and executing a 15x15 cm craniotomy with a "C-shape" durotomy. Dural closure will be at the discretion of the surgeon and the availability of resources, including duroplasty with aponeurotic galea, a suturable dural patch, a non-suturable dural patch, or simply a superficial dural cover with hemostatic materials like Surgicel® or Gelfoam®.

The expansion craniotomy will be finished with a cranioplasty using specific mini plates (3-5 "Rialto" plates) for bone fixation.

There are multiple techniques for DC. The elected technique will be at the discretion of the treating neurosurgeon, but only frontal-parietal-temporal DC will be considered. The removed bone flap may be stored in an abdominal pouch in the right or left upper abdominal quadrants or by freezing in a bone or blood bank freezer. Patients who receive an EC may subsequently be taken to DC if the expected improvement is not achieved with the intervention, according to the postsurgical images and invasive and noninvasive neuromonitoring, based on the criteria of the treating neurosurgeon. If this happens, the treating neurosurgeon must specify why they opted for the procedure. On the other hand, the intervention cannot be changed in patients taken to DC once the surgery is completed since the bone would have already been removed and stored.

ELIGIBILITY:
Inclusion Criteria:

1. TBI patients arriving at the emergency room in the first 24 hours following trauma.
2. Abnormal computed tomography (CT), with a primary injury including any epidural, intracerebral, or subdural collection with a midline shift >3mm and any basal cistern compression with at least 2 abnormal findings in the initial evaluation at the emergency room (including optic nerve ultrasound > 6mm at the same side of the CT´s primary injury or and/or an abnormal pupillometry with a reduced (Maximum Contraction Velocity) MCV in the pupil of the same side of the CT´s primary injury, or/and a Trans- Cranial Doppler (TCD) with Pulsatility Index (PI) > 1.3 and/or Middle Cerebral Artery - Diastolic Velocity (MCA-DV) < 20cm/seg on the same side of the CT´s primary injury or/and an Intracranial Pressure Pulse Wave (ICPPW) ICPPW2 > ICPPW1 waveform pattern in the same side of the CT´s primary injury).
3. Age 18 to 70 years old.
4. Patients with or without polytrauma with survival expectancy >24 hours.
5. Cranial decompression or cranial expansion surgical procedures less than 24 hours after the trauma.

Exclusion Criteria:

1. TBI patients arriving at the emergency room after 24 hours following trauma.
2. Normal CT scan at the emergency room.
3. Abnormal CT scan at the emergency room with any primary injury and midline shift less than 3mm or without basal cistern compression and with normal values in at least two different modalities of assessing ICCS (pupillometry, optic nerve sheath ultrasound, transcranial Doppler and/or non-invasive ICP waveform analyzer).
4. Age less than 18 or more than 70 years old.
5. Polytrauma or massive brain injury with survival expectancy < 24 hours.
6. Cranial decompression or cranial expansion surgical procedures performed > 24 hours after the trauma.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients arriving at any of the recruitment centers (tertiary hospitals or level 1 hospitals / specialized hospitals) in any of the involved countries (Bolivia, Brazil, Cambodia, Cameroon, Chile, Colombia, Dominican Republic, Ecuador, Egypt, Guatemala, Italy, Nigeria, Paraguay, Peru, Philippines, Rwanda, Serbia, Tanzania, Thailand, Venezuela).
Sampling Method: Non-Probability Sample
Enrollment: 292 (Estimated)
Dates: Start 2025-07-08 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
GOSE | Glasgow Outcome Scale Extended in different periods during one year
  Standard GOSE Evaluation without dichotomization.

SECONDARY OUTCOMES:
Surgical Site Complications | 1 year
  Post-operative CSF disturbances, surgical site infection, wound complications, number of required re-interventions.

OTHER OUTCOMES:
Post Operative Compliance Preservation | 15 days
  Control of the Intracranial Compartment Syndrome measured using ICP waveform via invasive and noninvasive devices and/or noninvasive neuromonitoring techniques (digital pupillometry, optic nerve sheath diameter ultrasonographic measurement, and transcranial Doppler) measured daily since ICU admission
Hospital Lenght of stay | 1 year
  ICU and in-hospital length of stay collected from medical records at hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Andres M Rubiano, MD, Principal Investigator — Meditech Foundation; Luigi V Berra, MD, Principal Investigator — La Sapienza University

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated during and/or analyzed during the current study will be available upon request to the key personnel of the sponsor institution. Individual participant data (IPD) will be stored in a private repository and made available upon request. Once requested, the unprocessed data collected on the RedCap platform will be shared as soon as possible. The shared data will be anonymous, as the only identifier will be the ID assigned to patients participating in the study. No additional consents are required for sharing IPD, as this possibility is included in the informed consent.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: From June 2025 to June 2027
Access Criteria: The datasets generated during and/or analyzed during the current study will be available upon request to the key personnel of the sponsor institution (see contact information). Individual participant data (IPD) will be stored in a private repository and made available upon request. Once requested, the unprocessed data collected on the RedCap platform will be shared as soon as possible. The shared data will be anonymous, as the only identifier will be the ID assigned to patients participating in the study. No additional consents are required for sharing IPD, as this possibility is included in the informed consent.
URL: http://www.space-tbi-study.com

REFERENCES:
- [Background] Berra LV, Cedrone G, Di Norcia V, D'Angelo L, Brunetto F, Familiari P, Palmieri M, Capobianco M, Pappone F, Santoro A. Development of a Novel Device for Decompressive Craniectomy: An Experimental and Cadaveric Study and Preliminary Clinical Application. Oper Neurosurg. 2023 Mar 1;24(3):324-330. doi: 10.1227/ons.0000000000000530. Epub 2022 Dec 12. PMID 36701747
- [Background] Godoy DA, Brasil S, Rubiano AM. Further support for the intracranial compartmental syndrome concept. Crit Care. 2024 Sep 18;28(1):311. doi: 10.1186/s13054-024-04974-4. No abstract available. PMID 39294706
- [Background] Palavani LB, Alves Neto LB, Batista S, Ferreira MY, Emmily de Carvalho D, de Vasconcellos Piscoya G, Teodoro Ramos Cabral Angelim Frazao C, Alves Leite JG, Fernandes MQ, Vieira Nogueira B, Godoy DA, Brasil S, Rubiano AM, Bertani de Magalhaes R, Paiva WS. Invasive and Noninvasive Techniques for Intracranial Pressure Monitoring After Decompressive Craniectomy: A Systematic Review and Meta-Analysis. World Neurosurg. 2024 Oct;190:76-87. doi: 10.1016/j.wneu.2024.06.118. Epub 2024 Jun 29. PMID 38950649
- [Background] Martinez-Palacios K, Vasquez-Garcia S, Fariyike OA, Robba C, Rubiano AM; noninvasive intracranial pressure monitoring international consensus group. Quantitative Pupillometry for Intracranial Pressure (ICP) Monitoring in Traumatic Brain Injury: A Scoping Review. Neurocrit Care. 2024 Aug;41(1):255-271. doi: 10.1007/s12028-023-01927-7. Epub 2024 Feb 13. PMID 38351298
- [Background] Martinez-Palacios K, Vasquez-Garcia S, Fariyike OA, Robba C, Rubiano AM; noninvasive ICP monitoring international consensus group. Using Optic Nerve Sheath Diameter for Intracranial Pressure (ICP) Monitoring in Traumatic Brain Injury: A Scoping Review. Neurocrit Care. 2024 Jun;40(3):1193-1212. doi: 10.1007/s12028-023-01884-1. Epub 2023 Dec 19. PMID 38114797
- [Background] Martinez-Palacios K, Vasquez-Garcia S, Fariyike OA, Robba C, Rubiano AM. Non-Invasive Methods for Intracranial Pressure Monitoring in Traumatic Brain Injury Using Transcranial Doppler: A Scoping Review. J Neurotrauma. 2024 Jun;41(11-12):1282-1298. doi: 10.1089/neu.2023.0001. Epub 2024 Apr 11. PMID 37861291
- [Background] Godoy DA, Brasil S, Iaccarino C, Paiva W, Rubiano AM. The intracranial compartmental syndrome: a proposed model for acute brain injury monitoring and management. Crit Care. 2023 Apr 10;27(1):137. doi: 10.1186/s13054-023-04427-4. PMID 37038236
- [Background] Rubiano AM, Figaji A, Hawryluk GW. Intracranial pressure management: moving beyond guidelines. Curr Opin Crit Care. 2022 Apr 1;28(2):101-110. doi: 10.1097/MCC.0000000000000920. PMID 35058406
- [Background] Mohan M, Layard Horsfall H, Solla DJF, Robertson FC, Adeleye AO, Teklemariam TL, Khan MM, Servadei F, Khan T, Karekezi C, Rubiano AM, Hutchinson PJ, Paiva WS, Kolias AG, Devi BI; NIHR Global Health Research Group on Neurotrauma. Decompressive craniotomy: an international survey of practice. Acta Neurochir (Wien). 2021 May;163(5):1415-1422. doi: 10.1007/s00701-021-04783-6. Epub 2021 Mar 18. PMID 33738561
- [Background] Iaccarino C, Kolias A, Adelson PD, Rubiano AM, Viaroli E, Buki A, Cinalli G, Fountas K, Khan T, Signoretti S, Waran V, Adeleye AO, Amorim R, Bertuccio A, Cama A, Chesnut RM, De Bonis P, Estraneo A, Figaji A, Florian SI, Formisano R, Frassanito P, Gatos C, Germano A, Giussani C, Hossain I, Kasprzak P, La Porta F, Lindner D, Maas AIR, Paiva W, Palma P, Park KB, Peretta P, Pompucci A, Posti J, Sengupta SK, Sinha A, Sinha V, Stefini R, Talamonti G, Tasiou A, Zona G, Zucchelli M, Hutchinson PJ, Servadei F. Consensus statement from the international consensus meeting on post-traumatic cranioplasty. Acta Neurochir (Wien). 2021 Feb;163(2):423-440. doi: 10.1007/s00701-020-04663-5. Epub 2020 Dec 22. PMID 33354733
- [Background] Hawryluk GWJ, Rubiano AM, Totten AM, O'Reilly C, Ullman JS, Bratton SL, Chesnut R, Harris OA, Kissoon N, Shutter L, Tasker RC, Vavilala MS, Wilberger J, Wright DW, Lumba-Brown A, Ghajar J. Guidelines for the Management of Severe Traumatic Brain Injury: 2020 Update of the Decompressive Craniectomy Recommendations. Neurosurgery. 2020 Sep 1;87(3):427-434. doi: 10.1093/neuros/nyaa278. PMID 32761068
- [Background] Layard Horsfall H, Mohan M, Devi BI, Adeleye AO, Shukla DP, Bhat D, Khan M, Clark DJ, Chari A, Servadei F, Khan T, Rubiano AM, Hutchinson PJ, Kolias AG. Hinge/floating craniotomy as an alternative technique for cerebral decompression: a scoping review. Neurosurg Rev. 2020 Dec;43(6):1493-1507. doi: 10.1007/s10143-019-01180-7. Epub 2019 Nov 11. PMID 31712994
- [Background] Hutchinson PJ, Kolias AG, Tajsic T, Adeleye A, Aklilu AT, Apriawan T, Bajamal AH, Barthelemy EJ, Devi BI, Bhat D, Bulters D, Chesnut R, Citerio G, Cooper DJ, Czosnyka M, Edem I, El-Ghandour NMF, Figaji A, Fountas KN, Gallagher C, Hawryluk GWJ, Iaccarino C, Joseph M, Khan T, Laeke T, Levchenko O, Liu B, Liu W, Maas A, Manley GT, Manson P, Mazzeo AT, Menon DK, Michael DB, Muehlschlegel S, Okonkwo DO, Park KB, Rosenfeld JV, Rosseau G, Rubiano AM, Shabani HK, Stocchetti N, Timmons SD, Timofeev I, Uff C, Ullman JS, Valadka A, Waran V, Wells A, Wilson MH, Servadei F. Consensus statement from the International Consensus Meeting on the Role of Decompressive Craniectomy in the Management of Traumatic Brain Injury : Consensus statement. Acta Neurochir (Wien). 2019 Jul;161(7):1261-1274. doi: 10.1007/s00701-019-03936-y. Epub 2019 May 28. PMID 31134383
- [Background] Clavijo A, Khan AA, Mendoza J, Montenegro JH, Johnson ED, Adeleye AO, Rubiano AM. The Role of Decompressive Craniectomy in Limited Resource Environments. Front Neurol. 2019 Feb 26;10:112. doi: 10.3389/fneur.2019.00112. eCollection 2019. PMID 30863354
- [Background] Rubiano AM, Maldonado M, Montenegro J, Restrepo CM, Khan AA, Monteiro R, Faleiro RM, Carreno JN, Amorim R, Paiva W, Munoz E, Paranhos J, Soto A, Armonda R, Rosenfeld JV. The Evolving Concept of Damage Control in Neurotrauma: Application of Military Protocols in Civilian Settings with Limited Resources. World Neurosurg. 2019 May;125:e82-e93. doi: 10.1016/j.wneu.2019.01.005. Epub 2019 Jan 16. PMID 30659971
- See also: Study Web Site — https://space-tbi-study.com/